CLINICAL TRIAL: NCT01272219
Title: Effect of Liraglutide on Body Weight in Non-diabetic Obese Subjects or Overweight Subjects With Co-morbidities: A Randomised, Double-blind, Placebo Controlled, Parallel Group, Multi-centre, Multinational Trial With Stratification of Subject to Either 56 or 160 Weeks of Treatment Based on Pre-diabetes Status at Randomisation
Brief Title: Effect of Liraglutide on Body Weight in Non-diabetic Obese Subjects or Overweight Subjects With Co-morbidities: SCALE™ - Obesity and Pre-diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-1839; 2008-001049-24 (EudraCT Number); U1111-1118-7871 (Other: WHO)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Liraglutide 3.0mg (week0-56)/Liraglutide 3.0mg (week56-68) (Experimental)
  Interventions: Drug: liraglutide
- Liraglutide 3.0mg (week0-56)/Liraglutide Placebo (week56-68) (Experimental)
  Interventions: Drug: placebo
- Liraglutide Placebo, no Pre-diabetes (Placebo Comparator)
  Interventions: Drug: placebo
- Liraglutide 3.0mg, Pre-diabetes (Experimental)
  Interventions: Drug: liraglutide
- Liraglutide Placebo, Pre-diabetes (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Subject with no pre-diabetes at screening, receiving liraglutide 3.0 mg subcutaneous (under the skin) injection once daily for 56 weeks. Subjects completing 56 weeks are re-randomised to receive liraglutide 3.0 mg for 12 weeks (until week 68).
  Arms: Liraglutide 3.0mg (week0-56)/Liraglutide 3.0mg (week56-68)
Drug: placebo — Subject with no pre-diabetes at screening, receiving liraglutide 3.0 mg subcutaneous (under the skin) injection once daily for 56 weeks. Subjects completing 56 weeks are re-randomised to receive liraglutide placebo for 12 weeks (until week 68).
  Arms: Liraglutide 3.0mg (week0-56)/Liraglutide Placebo (week56-68); Liraglutide Placebo, no Pre-diabetes
Drug: liraglutide — Liraglutide 3.0 mg, subcutaneous (under the skin) injection once daily for 160 weeks.
  Arms: Liraglutide 3.0mg, Pre-diabetes
Drug: placebo — Liraglutide placebo, subcutaneous (under the skin) injection once daily for 160 weeks.
  Arms: Liraglutide Placebo, Pre-diabetes

SUMMARY:
This trial is conducted in Africa, Asia, Europe, Oceania, North America and South America.

The aim of this clinical trial is to evaluate the potential of liraglutide to induce and maintain weight loss over 56 weeks in obese subjects or overweight subjects with co-morbidities. Furthermore, the aim is to investigate the long term potential of liraglutide to delay the onset of type 2 diabetes in subjects diagnosed with pre-diabetes at baseline.

Based on body mass index (BMI) and pre-diabetes status, subjects will be randomised to either 68 weeks (56 weeks of randomised treatment followed by a 12 week re-randomised treatment period) or 160 weeks of treatment (160 week treatment will only be applicable to subjects with pre-diabetes status at baseline).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Body Mass Index (BMI) of 30.0 kg/m^2 or above
* Body Mass Index (BMI) of 27 kg/m^2 or above in the presence of co-morbidities of treated or untreated dyslipidemia and/or hypertension
* Stable body weight
* Preceding failed dietary effort

Exclusion Criteria:

* Known type 1 or type 2 diabetes
* Glycosylated haemoglobin (HbA1c) of 6.5 % or above (Screening visit 1) or FPG of 126 mg/dL (7 mmol/L) or above (Screening visit 2) or 2 hour post-challenge (OGTT) plasma glucose of 200 mg/dL (11.1 mmol/L) or above (Screening visit 2)
* Screening calcitonin of 50 ng/L or above
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC)
* Personal history of non-familial medullary thyroid carcinoma
* History of acute or chronic pancreatitis
* Obesity induced by drug treatment
* Use of approved weight lowering pharmacotherapy
* Previous surgical treatment of obesity
* History of major depressive disorder or suicide attempt
* Uncontrolled hypertension (systolic blood pressure of 160 mmHg or above and/or diastolic blood pressure of 100 mmHg or above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3731 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2013-03-18 (Actual); Study Completion 2015-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry GCR, 1452, Study Director — Novo Nordisk A/S
Locations (195):
- United States (67):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Santa Monica, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, New London, Connecticut
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Crystal River, Florida
  - Novo Nordisk Investigational Site, Daytona Beach, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Ponte Vedra, Florida
  - Novo Nordisk Investigational Site, South Miami, Florida
  - Novo Nordisk Investigational Site, Athens, Georgia
  - Novo Nordisk Investigational Site, Dunwoody, Georgia
  - Novo Nordisk Investigational Site, Sandy Springs, Georgia
  - Novo Nordisk Investigational Site, Suwanee, Georgia
  - Novo Nordisk Investigational Site, Aurora, Illinois
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Baton Rouge, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Elkridge, Maryland
  - Novo Nordisk Investigational Site, North Dartmouth, Massachusetts
  - Novo Nordisk Investigational Site, City of Saint Peters, Missouri
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, Cary, North Carolina
  - Novo Nordisk Investigational Site, Raleigh, North Carolina
  - Novo Nordisk Investigational Site, Canal Fulton, Ohio
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Wadsworth, Ohio
  - Novo Nordisk Investigational Site, Tulsa, Oklahoma
  - Novo Nordisk Investigational Site, Eugene, Oregon
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, West Reading, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, West Jordan, Utah
  - Novo Nordisk Investigational Site, Arlington, Virginia
  - Novo Nordisk Investigational Site, Henrico, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Virginia Beach, Virginia
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Wenatchee, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Argentina (4):
  - Novo Nordisk Investigational Site, Ciudad Autónoma de Bs As
  - Novo Nordisk Investigational Site, Ciudad Autónoma de BsAs
  - Novo Nordisk Investigational Site, Ciudad de Buenos Aires
  - Novo Nordisk Investigational Site, Mar del Plata
- Australia (4):
  - Novo Nordisk Investigational Site, University of Sydney, New South Wales
  - Novo Nordisk Investigational Site, Woolloongabba, Queensland
  - Novo Nordisk Investigational Site, Adelaide, South Australia
  - Novo Nordisk Investigational Site, Heidelberg West, Victoria
- Austria (3):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Vienna
- Belgium (3):
  - Novo Nordisk Investigational Site, Boussu
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Liège
- Brazil (5):
  - Novo Nordisk Investigational Site, Porto Alegre, Rio Grande do Sul
  - Novo Nordisk Investigational Site, Campinas, São Paulo
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Curitiba
  - Novo Nordisk Investigational Site, São Paulo
- Canada (10):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Mount Pearl, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, St. John's, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Cambridge, Ontario
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Ottawa, Ontario
  - Novo Nordisk Investigational Site, Pointe-Claire, Quebec
  - Novo Nordisk Investigational Site, Québec
- Denmark (3):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Frederiksberg C
  - Novo Nordisk Investigational Site, Hvidovre
- Finland (3):
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, University of Helsinki
- France (5):
  - Novo Nordisk Investigational Site, Antibes
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Pierre-Bénite
  - Novo Nordisk Investigational Site, Saint-Herblain
- Germany (10):
  - Novo Nordisk Investigational Site, Bad Nauheim
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Freiburg im Breisgau
  - Novo Nordisk Investigational Site, Giessen
  - Novo Nordisk Investigational Site, Gifhorn
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Mannheim
  - Novo Nordisk Investigational Site, Saint Ingbert
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
- India (7):
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Belagavi, Karnataka
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Trichy, Tamil Nadu
  - Novo Nordisk Investigational Site, Karnāl
  - Novo Nordisk Investigational Site, Kerala
- Ireland (2):
  - Novo Nordisk Investigational Site, Dublin
  - Novo Nordisk Investigational Site, Galway
- Israel (7):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Ofakim
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Italy (8):
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Pisa
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Siena
- Mexico (6):
  - Novo Nordisk Investigational Site, Pachuca, Hidalgo
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Mexico City, México, D.F.
  - Novo Nordisk Investigational Site, Tampico, Tamaulipas
  - Novo Nordisk Investigational Site, Durango
  - Novo Nordisk Investigational Site, Monterrey
- Netherlands (7):
  - Novo Nordisk Investigational Site, Almere Stad
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Beek
  - Novo Nordisk Investigational Site, Hengelo OV
  - Novo Nordisk Investigational Site, Hilversum
  - Novo Nordisk Investigational Site, Leidschendam
  - Novo Nordisk Investigational Site, Zwijndrecht
- Norway (4):
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Trondheim
  - Novo Nordisk Investigational Site, Tønsberg
- Poland (5):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Katowice
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
- Russia (4):
  - Novo Nordisk Investigational Site, Arkhangelsk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Tyumen
- Novo Nordisk Investigational Site, Belgrade, Serbia and Montenegro
- Novo Nordisk Investigational Site, Belgrade, Serbia
- South Africa (3):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- Spain (6):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Santiago de Compostela
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valladolid
- Switzerland (5):
  - Novo Nordisk Investigational Site, Bern
  - Novo Nordisk Investigational Site, Dättwil
  - Novo Nordisk Investigational Site, Geneva
  - Novo Nordisk Investigational Site, Sankt Gallen
  - Novo Nordisk Investigational Site, Zollikerberg
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Istanbul
- United Kingdom (7):
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Luton
  - Novo Nordisk Investigational Site, Swansea

REFERENCES:
- [Result] Kolotkin RL, Fujioka K, Wolden ML, Brett JH, Bjorner JB. Improvements in health-related quality of life with liraglutide 3.0 mg compared with placebo in weight management. Clin Obes. 2016 Aug;6(4):233-42. doi: 10.1111/cob.12146. Epub 2016 May 19. PMID 27198973
- [Result] Overgaard RV, Petri KC, Jacobsen LV, Jensen CB. Liraglutide 3.0 mg for Weight Management: A Population Pharmacokinetic Analysis. Clin Pharmacokinet. 2016 Nov;55(11):1413-1422. doi: 10.1007/s40262-016-0410-7. PMID 27193270
- [Result] O'Neil PM, Garvey WT, Gonzalez-Campoy JM, Mora P, Ortiz RV, Guerrero G, Claudius B, Pi-Sunyer X; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. EFFECTS OF LIRAGLUTIDE 3.0 MG ON WEIGHT AND RISK FACTORS IN HISPANIC VERSUS NON-HIPANIC POPULATIONS: SUBGROUP ANALYSIS FROM SCALE RANDOMIZED TRIALS. Endocr Pract. 2016 Nov;22(11):1277-1287. doi: 10.4158/EP151181.OR. Epub 2016 Aug 2. PMID 27482610
- [Result] Fujioka K, O'Neil PM, Davies M, Greenway F, C W Lau D, Claudius B, Skjoth TV, Bjorn Jensen C, P H Wilding J. Early Weight Loss with Liraglutide 3.0 mg Predicts 1-Year Weight Loss and is Associated with Improvements in Clinical Markers. Obesity (Silver Spring). 2016 Nov;24(11):2278-2288. doi: 10.1002/oby.21629. PMID 27804269
- [Result] Bays H, Pi-Sunyer X, Hemmingsson JU, Claudius B, Jensen CB, Van Gaal L. Liraglutide 3.0 mg for weight management: weight-loss dependent and independent effects. Curr Med Res Opin. 2017 Feb;33(2):225-229. doi: 10.1080/03007995.2016.1251892. Epub 2016 Nov 6. PMID 27817208
- [Result] Wilding JP, Overgaard RV, Jacobsen LV, Jensen CB, le Roux CW. Exposure-response analyses of liraglutide 3.0 mg for weight management. Diabetes Obes Metab. 2016 May;18(5):491-9. doi: 10.1111/dom.12639. Epub 2016 Mar 1. PMID 26833744
- [Result] Pi-Sunyer X, Astrup A, Fujioka K, Greenway F, Halpern A, Krempf M, Lau DC, le Roux CW, Violante Ortiz R, Jensen CB, Wilding JP; SCALE Obesity and Prediabetes NN8022-1839 Study Group. A Randomized, Controlled Trial of 3.0 mg of Liraglutide in Weight Management. N Engl J Med. 2015 Jul 2;373(1):11-22. doi: 10.1056/NEJMoa1411892. PMID 26132939
- [Result] McEvoy BW. Missing data in clinical trials for weight management. J Biopharm Stat. 2016;26(1):30-6. doi: 10.1080/10543406.2015.1094814. PMID 26418188
- [Result] Ard J, Cannon A, Lewis CE, Lofton H, Vang Skjoth T, Stevenin B, Pi-Sunyer X. Efficacy and safety of liraglutide 3.0 mg for weight management are similar across races: subgroup analysis across the SCALE and phase II randomized trials. Diabetes Obes Metab. 2016 Apr;18(4):430-5. doi: 10.1111/dom.12632. Epub 2016 Feb 11. PMID 26744025
- [Result] le Roux CW, Astrup A, Fujioka K, Greenway F, Lau DCW, Van Gaal L, Ortiz RV, Wilding JPH, Skjoth TV, Manning LS, Pi-Sunyer X; SCALE Obesity Prediabetes NN8022-1839 Study Group. 3 years of liraglutide versus placebo for type 2 diabetes risk reduction and weight management in individuals with prediabetes: a randomised, double-blind trial. Lancet. 2017 Apr 8;389(10077):1399-1409. doi: 10.1016/S0140-6736(17)30069-7. Epub 2017 Feb 23. PMID 28237263
- [Result] von Scholten BJ, Davies MJ, Persson F, Hansen TW, Madsbad S, Endahl L, Jepsen CH, Rossing P. Effect of weight reductions on estimated kidney function: Post-hoc analysis of two randomized trials. J Diabetes Complications. 2017 Jul;31(7):1164-1168. doi: 10.1016/j.jdiacomp.2017.04.003. Epub 2017 Apr 11. PMID 28462892
- [Result] O'Neil PM, Aroda VR, Astrup A, Kushner R, Lau DCW, Wadden TA, Brett J, Cancino AP, Wilding JPH; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. Neuropsychiatric safety with liraglutide 3.0 mg for weight management: Results from randomized controlled phase 2 and 3a trials. Diabetes Obes Metab. 2017 Nov;19(11):1529-1536. doi: 10.1111/dom.12963. Epub 2017 Jul 21. PMID 28386912
- [Result] Davies MJ, Aronne LJ, Caterson ID, Thomsen AB, Jacobsen PB, Marso SP; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. Liraglutide and cardiovascular outcomes in adults with overweight or obesity: A post hoc analysis from SCALE randomized controlled trials. Diabetes Obes Metab. 2018 Mar;20(3):734-739. doi: 10.1111/dom.13125. Epub 2017 Nov 1. PMID 28950422
- [Result] Kolotkin RL, Gabriel Smolarz B, Meincke HH, Fujioka K. Improvements in health-related quality of life over 3 years with liraglutide 3.0 mg compared with placebo in participants with overweight or obesity. Clin Obes. 2018 Feb;8(1):1-10. doi: 10.1111/cob.12226. Epub 2017 Oct 16. PMID 29045079
- [Result] le Roux C, Aroda V, Hemmingsson J, Cancino AP, Christensen R, Pi-Sunyer X. Comparison of Efficacy and Safety of Liraglutide 3.0 mg in Individuals with BMI above and below 35 kg/m(2): A Post-hoc Analysis. Obes Facts. 2017;10(6):531-544. doi: 10.1159/000478099. Epub 2017 Nov 17. PMID 29145215
- [Derived] Kral P, Holst-Hansen T, Olivieri AV, Ivanescu C, Lamotte M, Larsen S. The Correlation Between Body Mass Index and Health-Related Quality of Life: Data from Two Weight Loss Intervention Studies. Adv Ther. 2024 Nov;41(11):4228-4247. doi: 10.1007/s12325-024-02932-8. Epub 2024 Sep 24. PMID 39316288
- [Derived] Williams DM, Staff M, Bain SC, Min T. Glucagon-like Peptide-1 Receptor Analogues for the Treatment of Obesity. touchREV Endocrinol. 2022 Mar;18(1):43-48. doi: 10.17925/EE.2022.18.1.43. Epub 2022 Mar 18. PMID 35975210
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 191 sites in 27 countries: Australia:4,Austria:3,Belgium:2, Brazil:5,Canada:11, Denmark:3,Finland:3, France:5, Germany:8,Hong Kong:1, Hungary:2, India:8, Ireland:1,Israel:7, Italy:7, Mexico:4, Netherlands:5, Norway:3, Poland:5, Russian:7, Serbia:2, South Africa:3, Spain:6, Switzerland:5,Turkey:4, UK:8, US:69.
Pre-assignment Details: Subjects were stratified based on pre-diabetes status and BMI at screening. The Main Period table, below, reflects the stratification that should have occurred at baseline. The Re-randomized Period and Main + Extension Period tables reflect the actual distribution of subjects, factoring in an incorrect stratification of 43 subjects at screening.
Groups:
- Liraglutide 3.0 mg, no Pre-diabetes: Arm 1 (Arm 1A + Arm 1B): Subjects with no pre-diabetes at screening received liraglutide 3.0 mg, once daily (OD) subcutaneously (s.c. injection, under the skin) for 56 weeks followed by a re-randomisation (1:1 into liraglutide 3.0 mg or liraglutide placebo) period of 12 weeks (weeks 56-68) and then an off-drug follow-up period of 2 weeks. The total duration of this treatment arm from randomisation to follow-up was 70 weeks.
- Liraglutide 3.0mg (week0-56)/Liraglutide 3.0mg (week56-68): Arm 1A: Subjects of Arm 1 (with no pre-diabetes at screening) receiving liraglutide 3.0 mg, once daily (OD) subcutaneously (s.c. injection, under the skin) for 56 weeks were re-randomised (1:1 into liraglutide 3.0 mg or liraglutide placebo) to continue treatment with liraglutide 3.0 mg for the next 12 weeks (weeks 56-68), followed by a 2 weeks off-drug follow-up period.
- Liraglutide 3.0mg (week0-56)/Liraglutide Placebo (week56-68): Arm 1B: Subjects of Arm 1 (with no pre-diabetes at screening) receiving liraglutide 3.0 mg, once daily (OD) subcutaneously (s.c. injection, under the skin) for 56 weeks were re-randomised (1:1 into liraglutide 3.0 mg or liraglutide placebo) to receive liraglutide placebo for the next 12 weeks (weeks 56-68), followed by a 2 weeks off-drug follow-up period.
- Liraglutide Placebo, no Pre-diabetes: Arm 2: Subjects with no pre-diabetes at screening received liraglutide placebo once daily (OD) subcutaneously (s.c. injection, under the skin) for 56 weeks and then continued with liraglutide placebo for additional 12 weeks (weeks 56-68), followed by a 2 weeks off-drug follow-up period. The total duration of this treatment arm from randomisation to follow-up was 70 weeks.
- Liraglutide 3.0 mg, Pre-diabetes: Arm 3: Subjects with pre-diabetes at screening received liraglutide 3.0 mg, once daily (OD) subcutaneously (s.c. injection, under the skin) for initial 56 weeks then continued treatment till 160 weeks, followed by an off-drug, observational follow-up period of 12 weeks. The total duration of this treatment arm from randomisation to follow-up was 172 weeks.
- Liraglutide Placebo, Pre-diabetes: Arm 4: Subjects with pre-diabetes at screening received liraglutide placebo once daily (OD) subcutaneously (s.c. injection, under the skin) for initial 56 weeks then continued treatment till 160 weeks, followed by an off-drug, observational follow-up period of 12 weeks. The total duration of this treatment arm from randomisation to follow-up was 172 weeks.
Period: Main Period: Week 0 to Week 56
Arm/Group | Liraglutide 3.0 mg, no Pre-diabetes | Liraglutide 3.0mg (week0-56)/Liraglutide 3.0mg (week56-68) | Liraglutide 3.0mg (week0-56)/Liraglutide Placebo (week56-68) | Liraglutide Placebo, no Pre-diabetes | Liraglutide 3.0 mg, Pre-diabetes | Liraglutide Placebo, Pre-diabetes
Started | 959 | 0 (This arm is not considered for main period as these subjects belong to re-randomised period) | 0 (This arm is not considered for main period as these subjects belong to re-randomised period) | 487 | 1528 | 757
Exposed | 957 | 0 | 0 | 487 | 1524 | 755
Completed | 679 | 0 | 0 | 296 | 1110 | 505
Not Completed | 280 | 0 | 0 | 191 | 418 | 252
Not completed — Adverse Event | 86 | 0 | 0 | 16 | 152 | 29
Not completed — Lack of Efficacy | 11 | 0 | 0 | 14 | 12 | 22
Not completed — Protocol Violation | 25 | 0 | 0 | 18 | 40 | 20
Not completed — Withdrawal criteria | 122 | 0 | 0 | 114 | 172 | 147
Not completed — Unclassified | 36 | 0 | 0 | 29 | 42 | 34
Period: Re-randomised Period: Week 56 to Week 68
Arm/Group | Liraglutide 3.0 mg, no Pre-diabetes | Liraglutide 3.0mg (week0-56)/Liraglutide 3.0mg (week56-68) | Liraglutide 3.0mg (week0-56)/Liraglutide Placebo (week56-68) | Liraglutide Placebo, no Pre-diabetes | Liraglutide 3.0 mg, Pre-diabetes | Liraglutide Placebo, Pre-diabetes
Started | 0 (This arm is not considered for re-randomised period as these subjects belong to main period) | 351 (Incorrect stratification: In this period, overall 37 pre-diabetic subjects were included by error.) | 350 (Incorrect stratification: In this period, overall 37 pre-diabetic subjects were included by error.) | 304 (Incorrect stratification: In this period, overall 37 pre-diabetic subjects were included by error.) | 0 (This arm is not considered for re-randomised period as these subjects belong to main period) | 0 (This arm is not considered for re-randomised period as these subjects belong to main period)
Completed | 0 | 342 | 343 | 289 | 0 | 0
Not Completed | 0 | 9 | 7 | 15 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 3 | 0 | 0
Not completed — Withdrawal criteria | 0 | 6 | 4 | 7 | 0 | 0
Not completed — Unclassified | 0 | 1 | 2 | 2 | 0 | 0
Period: Main + Extension Period: Week 0-172
Arm/Group | Liraglutide 3.0 mg, no Pre-diabetes | Liraglutide 3.0mg (week0-56)/Liraglutide 3.0mg (week56-68) | Liraglutide 3.0mg (week0-56)/Liraglutide Placebo (week56-68) | Liraglutide Placebo, no Pre-diabetes | Liraglutide 3.0 mg, Pre-diabetes | Liraglutide Placebo, Pre-diabetes
Started | 0 (This arm is not considered for this period as these subjects belong to main period) | 0 (This arm is not considered for this period as these subjects belong to re-randomised period) | 0 (This arm is not considered for this period as these subjects belong to re-randomised period) | 0 (This arm is not considered for this period as these subjects belong to main and re-randomised period) | 1505 (Incorrect stratification: In this period, overall 6 subjects with no pre-diabetes included by error.) | 749 (Incorrect stratification: In this period, overall 6 subjects with no pre-diabetes included by error.)
Exposed | 0 | 0 | 0 | 0 | 1501 | 747
Completed | 0 | 0 | 0 | 0 | 783 | 327
Not Completed | 0 | 0 | 0 | 0 | 722 | 422
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 191 | 43
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 29 | 36
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 76 | 36
Not completed — Withdrawal criteria | 0 | 0 | 0 | 0 | 364 | 256
Not completed — Missing reason | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Unclassified | 0 | 0 | 0 | 0 | 61 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide 3.0 mg, no Pre-diabetes | Liraglutide Placebo, no Pre-diabetes | Liraglutide 3.0 mg, Pre-diabetes | Liraglutide Placebo, Pre-diabetes | Total
Number analyzed (Participants) | 959 | 487 | 1528 | 757 | 3731
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (11.7) | 41.5 (11.5) | 47.4 (11.8) | 47.2 (11.8) | 45.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 801 | 390 | 1156 | 581 | 2928
  Male | 158 | 97 | 372 | 176 | 803
Fasting Body Weight [Mean (Standard Deviation); unit: kg] | 104.0 (20.1) | 103.6 (21.2) | 107.6 (21.8) | 107.9 (21.8) | 106.2 (21.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 37.5 (6.2) | 37.4 (6.2) | 38.8 (6.4) | 39.0 (6.3) | 38.3 (6.4)
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 5.3 (0.3) | 5.3 (0.3) | 5.8 (0.3) | 5.7 (0.3) | 5.6 (0.4)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 5.0 (0.4) | 5.1 (0.5) | 5.5 (0.6) | 5.5 (0.5) | 5.3 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fasting Body Weight
Description: The observed mean change from baseline in fasting body weight (%) after 56-weeks of treatment (main treatment period).
Time Frame: Week 0, Week 56
Population: The full analysis set (FAS) included all randomised subjects who were exposed to at least one dose of trial product (liraglutide 3.0 mg or liraglutide placebo) and who provided at least one post-baseline efficacy value. Missing data were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Liraglutide 3.0 mg (56-Week): Subjects belong to Arm 1 (with no pre-diabetes at screening) and Arm 3 (with pre-diabetes at screening), received liraglutide 3.0 mg, once daily (OD) subcutaneously (s.c. injection, under the skin) for 56 weeks, from randomisation.
- Liraglutide Placebo (56-Week): Subjects belong to Arm 2 (with no pre-diabetes at screening) and Arm 4 (with pre-diabetes at screening), received liraglutide Placebo, once daily (OD) subcutaneously (s.c. injection, under the skin) for 56 weeks, from randomisation.
Arm/Group | Liraglutide 3.0 mg (56-Week) | Liraglutide Placebo (56-Week)
Number analyzed (Participants) | 2432 | 1220
percent change | -7.98 (6.67) | -2.62 (5.74)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg (56-Week) vs Liraglutide Placebo (56-Week); Null-hypothesis: no treatment difference between treatment arms, i.e. liraglutide 3.0 mg and liraglutide placebo. Liraglutide 3.0 mg was considered superior to placebo in inducing and maintaining weight loss, if the estimated treatment effect (liraglutide 3.0 mg - liraglutide placebo) was statistically significantly smaller than zero; Test type: Superiority or Other; p < 0.0001, ANCOVA; Estimated mean difference = -5.39, 95% CI 2-sided [-5.82 to -4.95] — ANCOVA model with treatment, country, sex, pre-diabetes status at screening, baseline BMI stratum and an interaction between pre-diabetes status at screening and BMI stratum as fixed factors, and the baseline value as covariate

2. Primary Outcome: Proportion of Subjects Losing at Least 5% of Baseline Fasting Body Weight.
Description: Percentage of subjects losing at least 5% of baseline fasting body weight after 56-weeks of treatment (main treatment period).
Time Frame: At Week 56
Population: The FAS included all randomised subjects who were exposed to at least one dose of trial product (liraglutide 3.0 mg or liraglutide placebo) and who provided at least one post-baseline efficacy value. Missing data were imputed using LOCF.
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide 3.0 mg (56-Week) | Liraglutide Placebo (56-Week)
Number analyzed (Participants) | 2432 | 1220
percentage of subjects | 63.2 | 27.1
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg (56-Week) vs Liraglutide Placebo (56-Week); Null-hypothesis: no treatment difference between treatment arms, i.e. liraglutide 3.0 mg and liraglutide placebo. Liraglutide 3.0 mg was considered superior to placebo in inducing and maintaining weight loss as assessed by the proportion of subjects losing ≥5% of their fasting baseline weight, if the estimated odds ratio (liraglutide 3.0 mg/liraglutide placebo) was statistically significantly greater than one; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.80, 95% CI 2-sided [4.12 to 5.60] — The model included treatment, country, sex, pre-diabetes status at screening, BMI stratum and an interaction between pre-diabetes status at screening and BMI stratum as fixed factors, and the baseline value as covariate

3. Primary Outcome: Proportion of Subjects Losing More Than 10% of Baseline Fasting Body Weight
Description: Percentage of subjects losing >10% of baseline fasting body weight after 56-weeks of treatment (main treatment period).
Time Frame: At 56 weeks
Population: The FAS) included all randomised subjects who were exposed to at least one dose of trial product (liraglutide 3.0 mg or liraglutide placebo) and who provided at least one post-baseline efficacy value. Missing data were imputed using LOCF.
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide 3.0 mg (56-Week) | Liraglutide Placebo (56-Week)
Number analyzed (Participants) | 2432 | 1220
percentage of subjects | 33.1 | 10.6
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg (56-Week) vs Liraglutide Placebo (56-Week); Null-hypothesis: no treatment difference between treatment arms, i.e. liraglutide 3.0 mg and liraglutide placebo. Liraglutide 3.0 mg was considered superior to placebo in inducing and maintaining weight loss as assessed by the proportion of subjects losing >10% of their fasting baseline weight, if the estimated odds ratio (liraglutide 3.0 mg/liraglutide placebo) was statistically significantly greater than one; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.34, 95% CI 2-sided [3.54 to 5.32] — [estimate comment as in outcome 2, analysis 1]

4. Primary Outcome: Proportion of Subjects With Onset of Type 2 Diabetes
Description: Proportion of subjects with onset of Type 2 diabetes mellitus (T2DM) at week 160 (main + extension treatment period) among subjects with pre-diabetes at baseline - evaluated as time to onset of T2DM. Subjects included in FAS, who were stratified to 160-weeks of treatment (i.e., excluding 37 subjects with pre-diabetes who entered the re-randomised period and including 6 subjects without pre-diabetes incorrectly stratified to the 160-week treatment period).
Time Frame: At 160 weeks
Population: Subjects included in the FAS, who were stratified to 160-weeks of treatment; all randomised subjects who were exposed to at least one dose of trial product (liraglutide 3.0 mg or liraglutide placebo) and with at least one post-baseline efficacy measurement, who were stratified to 160-weeks of treatment. Missing data were imputed using LOCF.
Measure: Number; unit: Subject
Groups:
- Liraglutide 3.0 mg (160-Week): Subjects belong to Arm 3 (with pre-diabetes at screening), received liraglutide 3.0 mg, once daily (OD) subcutaneously (s.c. injection, under the skin) for 160 weeks, from randomisation.
- Liraglutide Placebo (160-Week): Subjects belong to Arm 4 (with pre-diabetes at screening), received liraglutide placebo, once daily (OD) subcutaneously (s.c. injection, under the skin) for 160 weeks, from randomisation.
Arm/Group | Liraglutide 3.0 mg (160-Week) | Liraglutide Placebo (160-Week)
Number analyzed (Participants) | 1472 | 738
Subject | 26 | 46
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg (160-Week) vs Liraglutide Placebo (160-Week); If the estimated time-to-event ratio (liraglutide 3.0 mg/ placebo), as assessed by the survival endpoint describing the time until onset of T2DM ('diabetes-free time'), is statistically significantly >1, then liraglutide 3.0 mg was to be considered superior to placebo in delaying the onset of T2DM in subjects with pre-diabetes at baseline. Weibull model was used; included treatment, sex and BMI stratification factor as fixed factors and baseline FPG as a covariate; Test type: Superiority or Other; p < .0001, Weibull analysis; Treatment estimate = 2.681, 95% CI 2-sided [1.856 to 3.872] — The treatment estimate was the factor that the time to event is multiplied with for liraglutide 3.0 mg compared to placebo

5. Secondary Outcome: Change From Baseline in Waist Circumference (cm)
Description: The observed mean change from baseline in waist circumference (cm) after 56-weeks of treatment (main treatment period).
Time Frame: Week 0, Week 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Liraglutide 3.0 mg (56-Week) | Liraglutide Placebo (56-Week)
Number analyzed (Participants) | 2437 | 1225
cm | -8.19 (7.31) | -3.94 (6.58)

6. Secondary Outcome: Change From Baseline in Waist Circumference (Subjects With Pre-diabetes at Baseline)
Description: The observed mean change from baseline in waist circumference (subjects with pre-diabetes at baseline) after 160 weeks of treatment (main + extension treatment period). Subjects included in FAS, who were stratified to 160-weeks of treatment (i.e., excluding 37 subjects with pre-diabetes who entered the re-randomised period and including 6 subjects without pre-diabetes incorrectly stratified to the 160-week treatment period).
Time Frame: Week 0, week 160
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Liraglutide 3.0 mg (160-Week) | Liraglutide Placebo (160-Week)
Number analyzed (Participants) | 1472 | 738
cm | -6.87 (8.28) | -3.37 (7.47)

7. Secondary Outcome: Pre-diabetes Status After 56 Weeks of Treatment
Description: Observed percentage of subjects with pre-diabetes status after 56 weeks of treatment (main treatment period).
Time Frame: Week 0, Week 56
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide 3.0 mg (56-Week) | Liraglutide Placebo (56-Week)
Number analyzed (Participants) | 2437 | 1225
percentage of subjects
  With No Pre-diabetes | 78.3 | 50.9
  With Pre-diabetes | 20.6 | 46.1
  With Transient Type 2 Diabetes | 0.9 | 1.8
  With Confirmed Type 2 Diabetes | 0.2 | 1.1

8. Secondary Outcome: Pre-diabetes Status in Subject With Pre-diabetes at Baseline After 160 Weeks of Treatment
Description: Observed percentage of subjects (subjects with pre-diabetes at baseline) with pre-diabetes status after 160 weeks of treatment (main + extension treatment period). Subjects included in FAS, who were stratified to 160-weeks of treatment (i.e., excluding 37 subjects with pre-diabetes who entered the re-randomised period and including 6 subjects without pre-diabetes incorrectly stratified to the 160-week treatment period).
Time Frame: Week 0, week 160
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide 3.0 mg (160-Week) | Liraglutide Placebo (160-Week)
Number analyzed (Participants) | 1472 | 738
percentage of subjects
  With No Pre-diabetes | 65.9 | 36.3
  With Pre-diabetes | 31.3 | 54.9
  With Transient Type 2 Diabetes | 1.1 | 2.6
  With Confirmed Type 2 Diabetes | 1.8 | 6.2

9. Secondary Outcome: Mean Change From Baseline in Fasting Body Weight (Subjects With Pre-diabetes at Baseline)
Description: The observed mean change from baseline in fasting body weight (subjects with pre-diabetes at baseline) after 160 weeks of treatment (main + extension treatment period). Subjects included in FAS, who were stratified to 160-weeks of treatment (i.e., excluding 37 subjects with pre-diabetes who entered the re-randomised period and including 6 subjects without pre-diabetes incorrectly stratified to the 160-week treatment period).
Time Frame: Week 0, week 160
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg (160-Week) | Liraglutide Placebo (160-Week)
Number analyzed (Participants) | 1467 | 734
percent change | -6.14 (7.34) | -1.89 (6.27)

10. Secondary Outcome: Proportion of Subjects Losing at Least 5% and Proportion of Subjects Losing More Than 10% of Baseline Fasting Body Weight (Subjects With Pre-diabetes at Baseline)
Description: Percentage of subjects losing >=5% and percentage of subjects losing >10% of baseline fasting body weight (pre-diabetic subjects at baseline) after 160-weeks of treatment (main + extension treatment period). Subjects included in FAS, who were stratified to 160-weeks of treatment (i.e., excluding 37 subjects with pre-diabetes who entered the re-randomised period and including 6 subjects without pre-diabetes incorrectly stratified to the 160-week treatment period).
Time Frame: At 160 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide 3.0 mg (160-Week) | Liraglutide Placebo (160-Week)
Number analyzed (Participants) | 1467 | 734
percentage of subjects
  Losing >=5% of baseline body weight | 49.6 | 23.7
  Losing >10% of baseline body weight | 24.8 | 9.9

11. Secondary Outcome: Change From Week 56 in Fasting Body Weight (%) (Re-randomised Subjects With No Pre-diabetes)
Description: The observed mean change in fasting body weight (%) from week 56 to week 68 in re-randomised subjects (with no pre-diabetes at baseline) after 12-weeks of treatment (re-randomised treatment period).
Time Frame: Week 56, Week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0mg (week0-56)/Liraglutide 3.0mg (week56-68) | Liraglutide 3.0mg (week0-56)/Liraglutide Placebo (week56-68) | Liraglutide Placebo, no Pre-diabetes
Number analyzed (Participants) | 349 | 346 | 299
percent change | 0.69 (2.58) | 2.91 (3.01) | 0.28 (2.39)

12. Secondary Outcome: Change From Baseline in Fasting Body Weight (%) (Re-randomised Subjects With No Pre-diabetes)
Description: The observed mean change from baseline in fasting body weight (%) in re-randomised subjects (with no pre-diabetes at baseline) after 68 weeks of treatment (main + re-randomised treatment period).
Time Frame: Week 0, Week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0mg (week0-56)/Liraglutide 3.0mg (week56-68) | Liraglutide 3.0mg (week0-56)/Liraglutide Placebo (week56-68) | Liraglutide Placebo, no Pre-diabetes
Number analyzed (Participants) | 349 | 347 | 298
percent change | -8.44 (7.23) | -6.77 (7.67) | -3.11 (7.52)

ADVERSE EVENTS:
Time Frame: For Arm 1 and Arm 2: week 0 to week 70 (68 weeks of treatment period + 2 weeks of follow-up). For Arm 3 and Arm 4: week 0 to week 172 (160 weeks of treatment period + 12 weeks of follow-up).
Description: A total of 37 pre-diabetic subjects erroneously entered the re randomised period and their adverse events (AEs) were counted under the "pre-diabetic arms" (Arm 3 and Arm 4). A total of 6 subjects without pre-diabetes incorrectly stratified to the 160-week treatment period and their AEs were counted under the "no pre-diabetes arms" (Arm 1 and Arm 2)
Arm/Group | Liraglutide 3.0 mg, Pre-diabetes | Liraglutide Placebo, Pre-diabetes | Liraglutide 3.0 mg, no Pre-diabetes | Liraglutide Placebo, no Pre-diabetes
Serious Adverse Events (participants affected / at risk) | 230/1524 | 96/755 | 59/957 | 19/487
Other Adverse Events (participants affected / at risk) | 1342/1524 | 586/755 | 843/957 | 345/487
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 3.0 mg, Pre-diabetes (N=1524) | Liraglutide Placebo, Pre-diabetes (N=755) | Liraglutide 3.0 mg, no Pre-diabetes (N=957) | Liraglutide Placebo, no Pre-diabetes (N=487)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bandaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple endocrine adenomatosis Type I (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basedow (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic nodular goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Barrett (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Caecitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Metaplasia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 6 (6) | 0 (0) | 2 (2) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 9 (9) | 1 (1) | 4 (4) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 22 (23) | 6 (6) | 7 (7) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amyloidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alveolar osteitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hepatitis A (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oophoritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug dispensing error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteric injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dupuytren (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 1 (1) | 0 (0)
Joint laxity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 (14) | 5 (6) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0) | 1 (1) | 2 (2)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mantle cell lymphoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord herniation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic adhesions (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polymenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cutis laxa (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excessive skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Miscarriage of partner (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominoplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart transplant (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mammoplasty (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Obesity surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectocele repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Varicophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 3.0 mg, Pre-diabetes (N=1524) | Liraglutide Placebo, Pre-diabetes (N=755) | Liraglutide 3.0 mg, no Pre-diabetes (N=957) | Liraglutide Placebo, no Pre-diabetes (N=487)
Abdominal pain (Gastrointestinal disorders) | 112 (150) | 37 (49) | 62 (79) | 19 (22)
Abdominal pain upper (Gastrointestinal disorders) | 110 (137) | 40 (49) | 63 (84) | 18 (20)
Constipation (Gastrointestinal disorders) | 333 (422) | 85 (100) | 203 (255) | 44 (52)
Diarrhoea (Gastrointestinal disorders) | 388 (626) | 107 (144) | 201 (308) | 46 (58)
Dyspepsia (Gastrointestinal disorders) | 156 (196) | 35 (40) | 102 (121) | 14 (16)
Eructation (Gastrointestinal disorders) | 86 (96) | 4 (4) | 38 (52) | 2 (2)
Flatulence (Gastrointestinal disorders) | 81 (94) | 22 (25) | 29 (35) | 15 (17)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 101 (112) | 18 (19) | 47 (50) | 8 (8)
Nausea (Gastrointestinal disorders) | 622 (974) | 128 (170) | 418 (616) | 78 (96)
Vomiting (Gastrointestinal disorders) | 300 (476) | 42 (55) | 172 (267) | 25 (29)
Fatigue (General disorders) | 154 (190) | 58 (67) | 79 (89) | 27 (31)
Injection site haematoma (General disorders) | 91 (102) | 61 (69) | 64 (68) | 42 (45)
Oedema peripheral (General disorders) | 53 (60) | 47 (58) | 22 (25) | 6 (7)
Bronchitis (Infections and infestations) | 114 (139) | 62 (80) | 35 (41) | 26 (27)
Gastroenteritis (Infections and infestations) | 138 (171) | 46 (53) | 48 (53) | 24 (32)
Influenza (Infections and infestations) | 181 (249) | 80 (123) | 65 (84) | 26 (37)
Nasopharyngitis (Infections and infestations) | 404 (764) | 210 (408) | 193 (290) | 110 (166)
Sinusitis (Infections and infestations) | 129 (174) | 65 (111) | 84 (99) | 35 (47)
Upper respiratory tract infection (Infections and infestations) | 236 (389) | 120 (213) | 101 (122) | 54 (68)
Urinary tract infection (Infections and infestations) | 123 (176) | 43 (62) | 48 (60) | 15 (19)
Lipase increased (Investigations) | 145 (207) | 24 (26) | 35 (41) | 10 (10)
Decreased appetite (Metabolism and nutrition disorders) | 169 (181) | 27 (28) | 102 (111) | 16 (17)
Hypoglycaemia (Metabolism and nutrition disorders) | 295 (637) | 35 (52) | 176 (302) | 29 (37)
Arthralgia (Musculoskeletal and connective tissue disorders) | 186 (231) | 97 (134) | 38 (41) | 23 (29)
Back pain (Musculoskeletal and connective tissue disorders) | 198 (283) | 118 (159) | 77 (97) | 41 (50)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 108 (127) | 54 (64) | 25 (27) | 22 (24)
Dizziness (Nervous system disorders) | 149 (197) | 55 (73) | 67 (81) | 19 (20)
Headache (Nervous system disorders) | 273 (432) | 124 (223) | 127 (178) | 58 (80)
Cough (Respiratory, thoracic and mediastinal disorders) | 112 (133) | 60 (87) | 34 (35) | 22 (23)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 74 (81) | 44 (52) | 31 (34) | 21 (22)
Hypertension (Vascular disorders) | 74 (86) | 48 (58) | 22 (23) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
When the primary results are available, Novo Nordisk plans to discuss the interpretation of these with the principal Investigator, but reserves the right to release results that may impact Novo Nordisk financial expectations (e.g. a press release directly to the public or similar) without prior consultation with the remaining participating Investigators. Novo Nordisk reserves the right not to release data until specified milestones, e.g. a clinical trial report is available.